CLINICAL TRIAL: NCT02198534
Title: Comparison of the Freiburg Visual Acuity Test (FrACT) With the EDTRS- and Landoltring Charts: a) Assessment of the Inter-test Agreement and the Test-retest Reliability b) Analysis of Examinees' / Examiner's Subjective Rating and of Test Durations
Brief Title: Comparison of the Freiburg Visual Acuity Test (FrACT) With the EDTRS- and Landoltring Charts
Acronym: FEL
Status: Completed | Type: Observational
Sponsor: Schiefer Ulrich (Other)
Responsible Party: Sponsor-Investigator, Schiefer Ulrich, Prof. Dr. med., Aalen University
Organization: Aalen University (Other)
Other Study IDs: F-2014-049
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Ophthalmologically Normal Subjects
Keywords: visual acuity; Landolt C; ETDRS charts; Freiburg Visual Acuity Test; FrACT; Comparison; acceptance; Test retest reliability; duration; questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — None applicable
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ophthalomogically normal subjects
  Interventions: Device: Methodology of visual acuity assessment

INTERVENTIONS:
Device: Methodology of visual acuity assessment
  Other Names: VISUCAT; FrACT; ETDRS Chart; Landolt C

SUMMARY:
A) For the investigation of Visual acuity, inter-test agreement and the test-retest reliability were used three different visual acuity tests: ETDRS charts, Landoltring chart and Freiburg Visual Acuity Test (FrACt). The examinees passed each visual acuity test twice but the sequence of the visual acuity tests were randomize and so different for each examinee. The examinees were 24 adult Aalen university students (except students of ophthalmic optics in terms 2 - 7) with a minimal distant visual acuity without or with correction of 0.2. Another inclusion criteria was a maximum myopia of sph -2,00 dpt, a maximum hyperopia of sph +5,50 dpt and a maximum astigmatism of cyl 2,50 dpt. The Landolt C was projected in eight-orientations. For the FrACT Test we used two different devices for response input: a modified keypad with Landoltring symbols (FrACTk) and a haptic Landolt device with an adjustable Landoltring (FrACTh). The primary objective was the comparison between FrACTk and FrACTh. The secondary Objective contains the comparison between all visual acuity tests.

B) Background: Landolt Cs and letters are commonly used optotypes. In the explorative study we compare four different ways of applying them: The Freiburg visual acuity test (FrACT) using a keypad and a haptic Landolt device, a Landolt C chart in accordance to ISO 8596 and DIN 58220 with eight-orientated Landolt C and ETDRS charts. The aims of the survey were to determine examinee´s/examiner´s subjective ratings using Visual analogue scales (VAS), the inter-test agreement between the tests and test-retest reliability of the tests, concerning the test duration.

Subjects and Methods: Twenty-four adult examinees with a visual acuity of ≥ 0,2 were included in the explorative study. The visual acuity of one eye was measured monocularly, randomized with regard to the leading/non-leading eye. The subjects passed every visual acuity test twice in a randomized sequence of the visual acuity tests, which is maintained by a pre-specified randomization list, making use of forced choice.

DETAILED DESCRIPTION:
1. FrACT (internet version 3.8.1) 1.1 haptic Landolt Ring device (FrACTh) 1.2 modified keypad with Landolt Ring symbols (FrACTk)
2. ETDRS Visual Acuity Tester (Steinbeis Transferzentrum Biomedizinische Optik, Tübingen/Germany)
3. Landoltring chart (Visus GmbH, Stuttgart/Germany)
4. VISUCAT monitor with single optotype display(numbers; Argus Individuell Optic GmbG, Putzbrunn/Germany)
5. Room illuminance level 250 lx, assessed with digital luxmeter (Peak Tech 5025, Peak Tech Prüf - und Messtechnik GmbH, Ahrensburg/Germany)
6. Laptopdisplay (TravelMate, Acer, 8372 Taipeh/China):

   luminance level 151 cd/m2 , surround luminance level 75 cd/m2 , assessed with luminance meter (IS-110 Laptop Minolta, Tokyo/Japan)
7. ETDRS Visual Acuity Tester:

   luminance level: 237 cd/m², surround luminance level 85 cd/m²
8. Landoltring Chart:

   luminance level: 236 cd/m², surround luminance level 84 cd/m²
9. VISUCAT:

   luminance level: 380 cd/m², surround luminance level 70 cd/m²
10. Stopwatch (Apple iPhone 4S, Cupertino CA/USA)
11. Laser Rangefinder (GLM 80 Professional, Bosch GmbH, Stuttgart/Germany)

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Minimum distant visual acuity (without/with correction) 0.2 (Visucat, single letter optotypes [numbers], initial session). As long as minimum distant visual acuity limits are exceeded, test runs without optical corrections are preferred in order to enhance the spectrum/variety of tested visual acuity values
* Ametropia:

maximum myopia sph -2.00 dpt maximum hyperopia sph +5.50 dpt maximum astigmatism cyl 2.5 dpt

* informed consent

Exclusion Criteria:

* Epilepsy / psychiatric disorders
* Drugs affect the reaction time and / or determining the visual acuity, or the refractive power of the eye
* Ophthalmic Education
* Amblyopia
* strabismus
* Glaucoma IOP> 22 mmHg
* Nystagmus
* Diabetic retinopathy (blood sugar-related retinal disease)
* Very dry eyes (sicca symptoms)
* eye surgery back are less than 3 months
* Infectious diseases (conjunctivitis, corneal inflammation, choroidal inflammation)
* miosis drugs
* Pronounced eye injuries
* Other eye disorders that affect the image quality
* Macular diseases
* albinism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmologically normal subjects
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
A) 1.Visual acuity (in terms of spatial resolution) | July - August, 2014 (1 month)
  Comparison of visual acuity measurements, visualized by Bland-Altman plots
Inter-test agreement between FrACTh and FrACTk with regard to visual acuity results | July - August, 2014 (1 month)
  Assessment of inter-test agreement between FrACTh and FrACTk by comparison between these two methods, visualized by Bland-Altman plots
Test-retest reliability of FrACTh and FrACTk with regard to visual acuity results | July - August, 2014 (1 month)
  Assessment of test-retest reliability of FrACTh and FrACTk by repeated measurements, visualized by Bland-Altman plots

SECONDARY OUTCOMES:
Examinees´ / examer's subjective ratings regarding the test procedures | July - August, 2014 (1 month)
  Assessment of examinees´ / examiner´s subjective ratings, using box & whisker plots for analysis of the visual analogue scale (VAS) results
Test duration (in seconds) | July - August, 2014 (1 month)
  Assessment of test duration and its comparison, using box & whisker plots and/or Bland-Altman plots

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof. Dr. med., Principal Investigator — University of Applied Sciences Aalen
Locations (1):
- University of Applied Sciences, Study Course Ophthalmic Optics, Aalen, Baden-Wurttemberg, Germany